CLINICAL TRIAL: NCT02513628
Title: The Optic Nerve Sheath Diameter for Prediction of Outcome After Cardiac Arrest: a Pilot Prospective Study
Brief Title: Optic Nerve Sheath Diameter for Prediction of Outcome After Cardiac Arrest
Acronym: ONSD-CA
Status: Completed | Type: Observational
Sponsor: Hopital of Melun (Other)
Responsible Party: Principal Investigator, Chelly Jonathan, MD, Hopital of Melun
Other Study IDs: MelunH
Record Dates: First submitted 2015-07-24; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; neuroprognostication; optic nerve sheath diameter; outcome; ultrasonography
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Early prognostication in resuscitated cardiac arrest (CA) patients, within the first day after admission in the intensive care unit (ICU), remains difficult. Optic nerve sheath diameter (ONSD) measurement could predict increased intracranial pressure. Preliminary works showed that ONSD measurement could be used to predict outcome in post-CA patients.

The aim of this study was to assess the ability of bedside ONSD ultrasonographic measurement to predict survival and Cerebral Performance Category (CPC) score at hospital discharge in post-cardiac arrest patients treated with therapeutic hypothermia (TH).

DETAILED DESCRIPTION:
Prospective observational study including all consecutive successfully resuscitated and TH-treated CA patients without traumatic or neurological etiology of CA in two French ICUs. ONSD measurements were performed on day 1, 2, and 3 after return of spontaneous circulation (ONSD1,2,3 respectively).

The primary outcome is survival at hospital discharge (with an average follow-up of 3 month until ICU admission).

ELIGIBILITY:
Inclusion Criteria:

* Unconscious (Glasgow Coma Scale ≤6)
* ≥18 years old
* Admitted in ICU after successful resuscitation from CA
* Treated with TH targeted to 33°C

Exclusion Criteria:

* unavailable ONSD measurement within 24 hours after return of spontaneous circulation (unavailable investigator, early death, or major hemodynamic instability)
* Traumatic or neurological origin of CA
* Previous cerebrovascular disease
* Facial trauma affecting the orbits and/or eyeballs
* Previous history of ocular pathology such as exophthalmia, glaucoma or cataract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All unconscious (Glasgow Coma Scale ≤6) patients ≥18 years old, admitted in ICU after successful resuscitation from CA, and treated with TH targeted to 33°C were screened. Exclusion criteria were as follows: unavailable ONSD measurement within 24 hours after return of spontaneous circulation (unavailable investigator, early death, or major hemodynamic instability), traumatic or neurological origin of CA, previous cerebrovascular disease, facial trauma affecting the orbits and/or eyeballs, and previous history of ocular pathology such as exophthalmia, glaucoma or cataract.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 3 months
  participants will be followed for the duration of hospital stay, an expected average of 3 months.